CLINICAL TRIAL: NCT06571916
Title: Investigating the Efficacy of a Novel Therapy for Suicide Risk in Adults: A Randomized Controlled Trial of an Intensive Single Session of "Brief Skills for Safer Living"
Brief Title: Brief Skills for Safer Living (Brief-SfSL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSL-02
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Suicide Prevention; Suicide; Suicide and Self-harm
Keywords: suicide; psychotherapy
MeSH Terms: conditions — Suicide Prevention; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief-SfSL (B-TAU) (Experimental): Participants will receive the Brief-SfSL treatment within 1 week of their screening.
  Interventions: Behavioral: Brief-SfSL
- Wait List (WL-TAU) (No Intervention): Participants will be put on a wait list and receive the Brief-SfSL treatment 3 months after their screening.

INTERVENTIONS:
Behavioral: Brief-SfSL — Brief-SfSL is a single 90-minute intervention that that:
  1. helps clients understand their suicide narrative, which explores the origin and meaning of their suicidal thoughts
  2. builds specific skills to keep oneself safe from suicide even if suicidal thoughts are present
  3. includes enhanced safety planning by identifying the barriers to enacting a safety plan and solutions to overcome them
  Other Names: Brief-Skills for Safer Living
  Arms: Brief-SfSL (B-TAU)

SUMMARY:
The goal of this project is to assess the efficacy of Brief-Skills for Safer Living (Brief-SfSL) in a randomized control trial. The investigators will be testing 150 participants Canada-wide, half of which will be randomized to receive Brief-SfSL (B-TAU) and the other half will be randomized to receive Brief-SfSL after a 3 month waitlist (WL-TAU). The main questions this study seeks to answer are:

* Is B-TAU more efficacious than WL-TAU for reducing suicidal thoughts at 3 months?
* Is B-TAU more efficacious than WL-TAU at 3 months for reducing depression severity, anxiety, and anhedonia?
* Is B-TAU more efficacious than WL-TAU at 3 months for improving social connectedness, emotional regulation, functioning (work, life, social), executive control and social problem-solving?
* Are adverse events equivalent between B-TAU and WL-TAU at 3 months?

DETAILED DESCRIPTION:
There are 2 million people in Canada at risk of death from suicide and suicide rates have not changed in the last 10 years. The COVID-19 pandemic also increased suicide risk and intensified a pre-existing lack of access to vital mental health services, with wait lists up to 1 year. To address this issue, the investigators developed "Brief Skills for Safer Living" (Brief-SfSL), a single-session individual psychotherapy intervention with the potential to make it easier to access care and shorten the time for people to access intervention. Derived from the proven success of the original SfSL 20-week group therapy, Brief-SfSL goes beyond conventional approaches by helping individuals understand their suicidal thoughts, build skills to manage these thoughts, and stay safe during crises. The strong results of the investigators single-arm trial of virtually-delivered Brief-SfSL in 77 adults with suicidal ideation across Canada show that Brief-SfSL is a feasible, acceptable, and safe intervention that has the potential to reduce suicide risk. To prove that it is, the investigators need to expand their study to include a treatment as usual (TAU) comparison group in a randomized controlled trial (RCT). The investigators will conduct an RCT that includes 2 groups: 75 participants who will receive TAU plus Brief-SfSL, and 75 who will receive TAU and be on a 3-month wait-list for Brief-SfSL. The aim is to compare the efficacy of Brief-SfSL vs. TAU on suicidal ideation and proxies for suicide risk (e.g., depression, anxiety) over 3 months. If the results confirm the efficacy of Brief-SfSL over TAU, this will provide definitive data to support the broad implementation of Brief-SfSL in hospitals and community mental health agencies across Canada. Study results will also be used to plan trials to assess the long-term impact of Brief-SfSL on suicide risk, healthcare system utilization, and health economics. Through this research, the investigators aim to save lives and also shift the paradigm of mental health intervention on a national scale.

ELIGIBILITY:
Inclusion Criteria:

* Suicidal ideation in the past week
* Access to a computer or phone with a camera
* Access to internet
* Access to an emergency contact and hospital within commuting distance
* Not receiving other psychotherapy/counselling services concurrently
* Willing to have the session recorded to determine therapy fidelity
* Any psychiatric diagnosis is allowed
* Follow-up visits with a psychiatrist and/or family doctor where a psychotherapeutic modality (e.g., Dialectical Behavioural Therapy, psychodynamic therapy, etc.) is not being used are allowable

Exclusion Criteria:

* Inability to undergo psychotherapy in English
* Presence of cognitive impairment that would limit consent and understanding of Brief Skills for Safer Living
* Active psychosis
* Unwilling or unable to provide informed consent
* Previously enrolled in the Brief-SfSL pilot study
* Unwilling or unable to communicate verbally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation using Beck Scale for Suicide Ideation | From baseline to 3 months post-intervention
  Beck Scale for Suicide Ideation is a 21-item self-report scale that quantifies suicidal ideation. Items are scored 0 to 2 and yield a total score ranging from 0 to 38. Higher scores reflect greater severity of suicidal ideation.

SECONDARY OUTCOMES:
Change in depression symptoms using the Quick Inventory of Depressive Symptoms 16-item scale (QIDS). | From baseline to 3 months post-intervention
  The QIDS is a 16-item validated depression scale. Total scores range from 0-27, with higher scores reflecting more severe depression.
Change in anxiety symptoms using the Generalized Anxiety Disorder 7-item scale (GAD-7) | From baseline to 3 months post-intervention
  The GAD-7 is a brief 7-item self-report scale measuring anxiety symptoms. Total scores range from 0 to 21, with higher scores reflecting more severe anxiety.
Changes in anhedonia using the Dimensional Anhedonia Rating Scale (DARS) | From baseline to 3 months post-intervention
  The DARS is a validated 17-item self-report scale measuring anhedonia across four domains. Total scores range from 0-68, with higher scores indicating lower levels of anhedonia.
Changes in feelings of social connectedness and burdensomeness using the Interpersonal Needs Questionnaire (INQ) | From baseline to 3 months post-intervention
  The INQ is a validated 15-item self-report scale assessing social connectedness and burdensomeness. Total scores range from 15-105, with higher scores indicating higher levels of social disconnectedness and burdensomeness.
Changes in work, social and family functioning using the Sheehan Disability Scale (SDS) | From baseline to 3 months post-intervention
  The SDS is a validated 3-item self-report scale that assesses work, social and family functioning. Total scores range from 0-30, with higher scores indicating higher impairment.
Changes in emotional dysregulation using the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) | From baseline to 3 months post-intervention
  The DERS-SF is an 18-item self-report scale that assesses emotional dysregulation across 6 subscales: (1) non-acceptance of emotional responses, (2) difficulties engaging in goal-directed behaviour, (3) impulse control difficulties, (4) lack of emotional awareness, (5) limited access to emotional regulation strategies and (6) lack of emotional clarity. Total scores range from 18-90, with higher scores reflecting more severe emotional dysregulation.
Changes in executive control using Space Explorer (gamified behavioural task) | From baseline to 3 months post-intervention
  The Space Explorer task is an Aversive Go/No-Go task that assesses active-escape biases or the reduced ability to withhold an escape response when exposed to an aversive context. The 2x2 factorial task design results in 4 different conditions, each associated with a distinct visual cue in the form of "space junk". The meanings of the cues are learned from experience across trials based on trial outcomes: neutral (e.g., silence, absence of any aversive/rewarding visual cues) or aversive/rewarding (e.g., aversive white noise, loss/gain of points, advancing in the game, etc.). Participants are naturally incentivized to try to maximize neutral/positive outcomes and avoid aversive outcomes by choosing the right action for a given cue: Go (pressing a button), or No-go (doing nothing and simply waiting). This task takes 10-15 minutes to complete.
Changes in social problem-solving using Jungle Treasure Hunt (gamified behavioural task) | From baseline to 3 months post-intervention
  The Jungle Treasure Hunt task tests players' ability to infer the intentions of others and adapt under uncertainty as they pursue rewarding outcomes. Players must navigate through a jungle and collect treasure by choosing between two paths on each trial. An avatar in the form of a monkey appears before each draw and recommends which path to take, with a speech bubble above the monkey stating "Choose the LEFT path" or "Choose the RIGHT path". The player then selects the left or right path and decides how many steps to take. The reward they receive is proportional to the number of steps they take, but if they choose the wrong path, they will lose rewards. The player's total score is shown and they are informed if they were correct or incorrect. Before the game starts, the player is told that the avatar's advice may not always be accurate. This task takes 15-20 minutes to complete.
Participant safety as measured by adverse events | Through study completion, an average of 3 months
  Participants will be asked to report any adverse events experienced at each visit. Investigators will measure if there are any differences in the number, severity or relatedness between group to ensure the intervention is safe.
Suicide severity differences between groups as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) | Through study completion, an average of 3 months
  The C-SSRS is a semi-structured clinical interview to assess suicidal ideation and behaviour (lifetime, current, and since last visit). Investigators will be analyzing if there is any difference in C-SSRS severity between groups to ensure safety of the intervention. Suicidal ideation is scored from 0-5, with 5 indicating greater severity. Intensity of suicidal ideation is scored from 0-5, with 5 indicating greater intensity. Lethality of actual suicide attempts is scored from 0-5, with 5 indicating greater lethality.

CONTACTS AND LOCATIONS:
Overall Officials: Sakina Rizvi, PhD, MACP, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No